CLINICAL TRIAL: NCT04999423
Title: Safety and Effectiveness Analysis of Stent Assisted Coiling With LVIS™ Evo™ and HydroCoil® Embolic System in Aneurysm Treatment
Brief Title: LVIS™ Evo™ and HydroCoil® Embolic System for Intracranial Aneurysm Treatment
Acronym: SEALANT
Status: Active, not recruiting | Type: Observational
Sponsor: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SEALANT
Record Dates: First submitted 2021-07-28; First posted 2021-08-10 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Intracranial Aneurysm
Keywords: aneurysm; endovascular; hydrocoil; stent assisted coiling; LVIS EVO
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: LVIS EVO and HydroCoil Embolic System — Stent assisted Coiling

SUMMARY:
This is a prospective multicenter international single-arm observational study to demonstrate that use of stent-assisted coiling with LVIS™ Evo™ and HydroCoil® Embolic System (HES) in intracranial aneurysm treatment is effective and safe when assessed at 1 year after the procedure

DETAILED DESCRIPTION:
Patient treatment and follow-up will be performed as per standard of care. The study will evaluate the proportion of aneurysms with complete occlusion based on Raymond-Roy occlusion classification (RROC) at 12 ± 6-months, as well as other effectiveness and safety endpoints such as the occurence of stent stenosis or parent artery occlusion, the occurence of retreatment and recanalization, the rate of major ipsilateral stroke or neurological death, the proportion of patients with good functional clinical outcome, the occurence of SAH, aneurysm rupture, procedural complications, serious adverse events...

Sample size: 200 patients

ELIGIBILITY:
Inclusion Criteria:

* IC 1. Patient whose age is 18 years old or above;
* IC 2. Patient (or legal representative, where applicable) who understands the study requirements and the treatment procedures and provides written informed consent before any study-specific procedures are performed;
* IC 3. Patient eligible for the treatment with LVIS™ Evo™ and HydroCoil® Embolic System (HES);
* IC 4. Patient whose target aneurysm is unruptured or ruptured (> 30 days since occurrence);
* IC 5. Patient whose target aneurysm size is less than or equal to 12 mm;
* IC 6. Patient willing to comply with all planned follow-ups and evaluations.

Exclusion Criteria:

* EC 1 Patient who has suffered an intracerebral hemorrhage within 30 days prior to the procedure;
* EC 2. Patient whose target aneurysm is a fusiform aneurysm;
* EC 3. Patient whose target aneurysm has previously been treated with a stent;
* EC 4. Patient whose target aneurysm is partially thrombosed;
* EC 5. Patient whose target aneurysm requires Y stenting;
* EC 6. Patient whose target aneurysm is associated with an arteriovenous malformation (cAVM), or any other lesion that could lead to hemorrhagic complications;
* EC 7. Patient who has more than one aneurysm to be treated during the same procedure, (except in case of an adjacent aneurysm that could be treated with the same stent);
* EC 8. Patient for whom the treatment with another stent than LVIS™ Evo™ or in addition to LVIS™ Evo™ is planned;
* EC 9. Patient with a planned treatment of other aneurysm in the same vascular territory within 12 months;
* EC 10. Patient who has a known allergy to contrast agents (that cannot be adequately premedicated) and/or to the study device or procedure-required concomitant medications or procedures (e.g. contraindication to antiplatelet and/or anticoagulants, allergy to Nickel-titanium or contraindication to MRI/MRA or angiography);
* EC 11. Patient who has one of the following (as assessed prior to the index procedure): Other serious medical illness (e.g., cancer or any severe or fatal comorbidity) with estimated life expectancy of less than the study duration, OR Planned procedure that may cause non-compliance with the protocol or confound data interpretation;
* EC 12. Patient who is participating or intends to participate in another study that changes the site practice (interventional) within the study time period;
* EC 13. Pregnant or breastfeeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with an unruptured or ruptured (> 30 days since occurrence) intracranial aneurysm eligible for endovascular treatment using LVIS™ Evo™ and HydroCoil® Embolic System (HES)
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of aneurysms with complete occlusion | 12 ± 6-month
  based on Raymond-Roy occlusion classification (RROC) evaluated by an independent Core laboratory using digital subtraction angiograms (DSA)

SECONDARY OUTCOMES:
Proportion of aneurysms with Raymond-Roy Occlusion Class I, II or III, and Modified Raymond-Roy Classification at immediate post procedure and each follow-up visits | 30 ± 6 months
  Raymond Roy Classification and Modified Raymond-Roy Classification evaluated by an independent Core laboratory
RROC shift between immediate post procedure and each follow-up visit | 30 ± 6 months
  based on Raymond Roy Classification evaluated by an independent Core laboratory
Aneurysm occlusion stability between immediate post procedure and each follow-up visit | 30 ± 6 months
  stable, improved, or worsened evaluated by an independent Core laboratory
Proportion of aneurysms with stent successful deployment at the target aneurysm neck | Day 0
  evaluated by an independent Core laboratory
Percentage of HES coil length implanted in the target aneurysm | Day 0
  HES coil length on the total coil length used
Proportion of aneurysms with complete stent apposition | Day 0
  evaluated by an independent Core laboratory
Occurrence of in-stent stenosis or parent artery occlusion at each follow-up | 30 ± 6 months
  evaluated by an independent Core laboratory
Occurrence of target aneurysm recanalization at each follow-up | 30 ± 6 months
  Aneurysm occlusion deterioration evaluated by an independent Core laboratory
Occurrence of target aneurysm retreatment at each follow-up | 30 ± 6 months
  Retreatment or planned retreatment
Major ipsilateral stroke or neurological death within 12 months and 30 months | 30 ± 6 months
  assessed by an independent clinical event committee
Proportion of patients with good functional clinical outcomes | 30 ± 6 months
  a good functional outcome is defined by an mRS between 0 and 2, or an mRS equal to baseline if it was > 2 at baseline, with mRS is the modified Rankin Scale (a neurological score from 0: no deficit to 6: death)
Occurrence of subarachnoid hemorrhage | 30 ± 6 months
  assessed by an independent clinical event committee
Occurrence of Aneurysm rupture | 30 ± 6 months
  assessed by an independent clinical event committee
Occurrence of device-related serious adverse events | 30 ± 6 months
  assessed by an independent clinical event committee
Occurrence of procedural complications | Day 0
  assessed by an independent clinical event committee
All-cause mortality rate | 30 ± 6 months
  assessed by an independent clinical event committee

CONTACTS AND LOCATIONS:
Overall Officials: Rene Chapot, Prof., Principal Investigator — Alfried Krupp Krankenhaus; Jonathan Downer, Dr., Principal Investigator — Royal Infirmary of Edinburgh
Locations (19):
- Charleroi University Hospital, Charleroi, Belgium
- France (6):
  - Brest University Hospital, Brest
  - Limoges University Hospital, Limoges
  - Lyon University Hospital, Lyon
  - Marseille University Hospital, Marseille
  - Fondation Rothschild, Paris
  - Rouen University Hospital, Rouen
- Germany (4):
  - Universitätsklinikum Augsburg, Augsburg
  - Universitätsklinikum Knappschaftskrankenhaus, Bochum
  - Alfried Krupp Krankenhaus, Essen
  - Universitätsklinikum Münster, Münster
- Italy (3):
  - Azienda Ospedaliera Cannizzaro, Catania
  - Policlinico Martino Messina, Messina
  - Ospedali riuniti San Giovanni di Dio e Ruggi d'Aragona, Salerno
- United Kingdom (5):
  - Royal Infirmary of Edinburgh, Edinburgh
  - Walton Centre, Liverpool
  - Charing Cross Hospital, London
  - King's College Hospital, London
  - The Royal London Hospital, London

IPD SHARING:
Plan to Share IPD: No